CLINICAL TRIAL: NCT01925040
Title: Clinical Investigation of a New Nanohybrid Resin Composite Venus Pearl in Class 2 Cavities- a Multi-center Study
Brief Title: Comparison of 2 Different Resin Based Filling Materials in Posterior Teeth - a Multicenter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heraeus Kulzer GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKG-DT-01/2011-SOCO-CLIN
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Caries; Unsatisfactory or Defective Restoration of Tooth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Venus Pearl (Experimental): Placement of restoration using Venus Pearl in carious teeth or as a replacement of a defective previous restoration.
  Interventions: Device: Placement of restoration
- control resin-based filling material (Active Comparator): Placement of restoration using a control resin-based filling material in carious teeth or as a replacement of a defective previous restoration.
  Interventions: Device: Placement of restoration

INTERVENTIONS:
Device: Placement of restoration — Placement of restorations

SUMMARY:
The purpose of this study is to compare the clinical performance of a new resin based filling material to an established resin-based filling material in posterior teeth at 2 different study centers.

DETAILED DESCRIPTION:
The objective of this study is to compare the performance of the composite resin Venus Pearl and a commercially available control composite material for the restoration of class II-cavities. Primary endpoints of the study are a mean score for each patient calculated from aesthetic, functional attribute and biological parameters. Secondary endpoints are the evaluation of secondary caries, plaque accumulation and gingival reactions and the comparison of the primary score at week 1, month 6, month 12 and month 24 after restoration. Beside this, the single components of the three categories of the primary endpoints will be compared. The study will be executed as a multi-center (Oregon Health & Science University, Portland, OR, USA and Medical School Hannover, Hannover, Germany), single-blinded and randomized clinical investigation. 90 comparable cavities per study site will be treated (45 cavities for each material at each site).

ELIGIBILITY:
Inclusion Criteria:

* Patients should be 18 years and older.
* Study teeth should have an interproximal (Class II) carious lesion or an existing defective class II restoration requiring restorative therapy on premolars or molars.
* The maximum cavity depth determined by the radiograph will be D2 (Tyas classification).
* The teeth included in the study need to have a proximal contact with the adjacent tooth and be in occlusion with the opposing dentition.
* The teeth included in the study should be vital with no signs of pulpal pathology.
* Patients that report brushing regularly without severe gingival inflammation and/or extensive caries.
* Patients should have no allergies or systemic diseases which inhibit the treatment.
* Patients should have voluntary participation and sign a written informed consent form.
* Patients should be willing to participate in the recall/re-examination appointments.

Exclusion Criteria:

* Simultaneous participation in another study about dental restorative materials.
* Written informed consent form not signed.
* Nonvital pulp / periapical lesion.
* Insufficient oral hygiene despite detailed instructions.
* Pregnancy/ breast feeding before placement of the study restoration.
* Minors.
* Severe malocclusion/ malalignment/ traumatic occlusion/ bruxism.
* Known allergy to any components present in any of the materials that are used for this study.
* Unclear mucosal alterations, e.g. oral lichenoid reactions/lesions.
* Severe medical complications (organ transplants, cancer, immune-compromised, long-term antibiotic or steroid therapy).
* Infectious diseases such as HIV/Aids, Hepatitis, etc.
* Application of bleaching products less than 14 days before placement of the restoration.
* Orthodontic treatment during the study.
* Xerostomia.
* Untreated periodontal diseases.
* Rampant or extensive caries present.
* Systemic diseases with potential oral manifestation.
* Sufficient isolation according to the criteria of adhesive techniques not possible, e.g. application of rubber dam.
* Direct adhesive restoration not indicated.
* Replacement of more than one cusp indicated.
* Dental fears patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Geurtsen, Prof. Dr., Study Chair — Hannover Medical School; Gabriela Ibarra, DDS, MPH, MS, Principal Investigator — Oregon Health and Science University; Werner Geurtsen, Prof. Dr., Principal Investigator — Medical School Hannover
Locations (2):
- Oregon Health and Science University-School of Dentistry, Portland, Oregon, United States
- Medical School Hannover, Hanover, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The total number of patients that started the study was 130. However, each patient was eligible to receive up to four restorations, with either a test or a control material. That means the same patient can have received a restoration/restorations with Venus Pearl as well as with the control resin-based filling material. That is the reason why the sum of the following participants differs from the total patient number 130. The analysis was restoration based.
Units Other Than Participants: restorations
Period: Overall Study
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Started | 85; 90 restorations (The total number of patients that started the study was 130. However, each patient was eligible to receive up to four restorations, with either a test or a control material. That means the same patient can have received a restoration/restorations with Venus Pearl as well as with the control resin-based filling material. That is the reason why the sum of the participants differs from the total patient number 130.) | 83; 90 restorations (The total number of patients that started the study was 130. However, each patient was eligible to receive up to four restorations, with either a test or a control material. That means the same patient can have received a restoration/restorations with Venus Pearl as well as with the control resin-based filling material. That is the reason why the sum of the participants differs from the total patient number 130.)
Completed | 49; 55 restorations | 48; 53 restorations
Not Completed | 36; 35 restorations | 35; 37 restorations

BASELINE CHARACTERISTICS:
Population: 90 restorations with each material were placed at T0 (in total 180). 7 days afterwards baseline analysis was performed and not all patients from T0 showed up at baseline. That is why the participant and restoration number between T0 and baseline differs.
  Each patient was eligible to receive up to 4 restorations, with either test or control material. That means the same patient can have received restoration(s)with VP as well as with control.116 is the absolute patient number at baseline.
Units Other Than Participants: Restorations
Groups:
- Total: Total of all reporting groups
Arm/Group | Venus Pearl | Control Resin-based Filling Material | Total
Number analyzed (Participants) | 78 | 75 | 116
Number analyzed (Restorations) | 83 | 80 | 163
Age, Customized [Number; unit: years] — Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  years
    < 18 years | 0 | 0 | 0
    18 - 75 years | 83 | 80 | 163
    > 75 years | 0 | 0 | 0
Sex: Female, Male [Count of Units; unit: Restorations] — Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  Restorations
    Female | 43 | 42 | 85
    Male | 40 | 38 | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Post-operative hypersensitivity [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.08 (0.28) | 1.06 (0.24) | 1.07 (0.26)
Caries, erosion [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.05 (0.22) | 1.06 (0.24) | 1.06 (0.25)
"Tooth integrity" [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.04 (0.19) | 1.06 (0.24) | 1.05 (0.22)
Parodontal reaction [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.17 (0.38) | 1.2 (0.51) | 1.18 (0.45)
Adjacent mucosa [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.12 (0.36) | 1.2 (0.49) | 1.16 (0.43)
Fracture and retention [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.10 (0.46) | 1.08 (0.31) | 1.09 (0.39)
Marginal adaptation [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.25 (0.58) | 1.16 (0.4) | 1.21 (0.5)
Abrasion [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.01 (0.11) | 1.03 (0.22) | 1.02 (0.17)
Approximal anatomical form [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.38 (0.7) | 1.29 (0.53) | 1.33 (0.62)
Surface luster [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.28 (0.51) | 1.28 (0.45) | 1.28 (0.48)
Satisfaction of patient [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.11 (0.44) | 1.06 (0.24) | 1.09 (0.36)
Marginal discoloration [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.16 (0.4) | 1.26 (0.5) | 1.18 (0.43)
Surface staining [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.11 (0.35) | 1.1 (0.3) | 1.1 (0.33)
Color match [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.27 (0.47) | 1.26 (0.5) | 1.26 (0.48)
Esthetic anatomical form [Mean (Standard Deviation); unit: scores on a scale] — 1. = Clinical excellent, very good
  2. = Clinically good
  3. = Clinically sufficient, satisfactory
  4. = Clinically unsatisfactory (reparable)
  5. = Clinically poor (replacement necessary) Population: Each patient was eligible to receive up to 4 restorations, with either VP or control. So, e.g. the same patient can have received 1 restoration with VP and 1 restoration with control. So, materialwise there is 1 patient for VP and 1 patient for control, which adds up in the ClinicalTrial system in the total column as 2 patients, even though it was only 1 patient. This is why the patient numbers in the columns do not represent the sum of the absolute patient number (116).
  scores on a scale | 1.22 (0.52) | 1.24 (0.48) | 1.22 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Score for Surface Luster
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of esthetic properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for surface luster
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.89 (0.6) | 1.62 (0.63)

2. Primary Outcome: Score for Surface Staining
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of esthetic properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for surface staining
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.44 (0.54) | 1.34 (0.52)

3. Primary Outcome: Score for Marginal Discoloration
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of esthetic properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for marginal discoloration
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.49 (0.57) | 1.47 (0.72)

4. Primary Outcome: Score for Fracture and Retention
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of functional properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for fracture and retention
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.24 (0.58) | 1.32 (0.64)

5. Primary Outcome: Score for Color Match
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of esthetic properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for color match
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.64 (0.7) | 1.64 (0.68)

6. Primary Outcome: Score for Esthetic Anatomical Form
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of esthetic properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for esthetic anatomical form
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.49 (0.63) | 1.45 (0.64)

7. Primary Outcome: Score for Marginal Adaptation
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of functional properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for marginal adaptation
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.29 (0.53) | 1.42 (0.69)

8. Primary Outcome: Score for Abrasion
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of functional properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for abrasion
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.16 (0.42) | 1.17 (0.43)

9. Primary Outcome: Score for Approximal Anatomical Form
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of functional properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for approximal anatomical form
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.44 (0.76) | 1.23 (0.51)

10. Primary Outcome: Score for Satisfaction of Patient
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of functional properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for satisfaction of patient
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.04 (0.27) | 1.06 (0.41)

11. Primary Outcome: Score for Post-operative Hypersensitivity
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of biological properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for post-operative hypersensitivity
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.04 (0.19) | 1.04 (0.19)

12. Primary Outcome: Score for Caries, Erosion
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of biological properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for caries, erosion
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.02 (0.13) | 1.08 (0.43)

13. Primary Outcome: Score for "Tooth Integrity"
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of biological properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for "tooth integrity"
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.11 (0.37) | 1.19 (0.44)

14. Primary Outcome: Score for Parodontal Reaction
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of biological properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for parodontal reaction
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.45 (0.77) | 1.36 (0.68)

15. Primary Outcome: Score for Adjacent Mucosa
Description: The primary endpoint will be a mean score calculated as following: There are three aspects to be assessed: aesthetic, functional attribute and biological parameters.
  Score of biological properties:
  1: Clinically excellent, 2: Clinically good, 3: Clinically sufficient, 4: Clinically unsatisfactory, 5: Clinically poor Score for adjacent mucosa
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Restorations
Arm/Group | Venus Pearl | Control Resin-based Filling Material
Number analyzed (Participants) | 55 | 53
Number analyzed (Restorations) | 55 | 53
scores on a scale | 1.07 (0.26) | 1.11 (0.42)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Venus Pearl | Control Resin-based Filling Material
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT01925040/Prot_SAP_000.pdf